CLINICAL TRIAL: NCT06913686
Title: Effect of Music on Mental and Physical Performance in Young Tennis Players : a Pre-experimental Study
Brief Title: Effect of Music on Mental and Physical Performance in Young Tennis Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Saoussen Layouni, Associate professor, Faculty of Medicine, Sousse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Department of physical medicin
Record Dates: First submitted 2025-03-25; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Physical Performances; Mental Performances
Keywords: Music; physical performance; mental training; ,stress management; concentration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Child and adolescents tennis players (Experimental): child and adolescent tennis players in the competitive category who are enrolled in the tennis club of La Marsa, Tunis in Tunisia and regularly engage in tennis practice.
  Interventions: Behavioral: Music intervention

INTERVENTIONS:
Behavioral: Music intervention — experimental controlled study will be conducted at the La Marsa tennis club in Tunis, Tunisia, utilizing a rigorous methodology to collect data from competitive young tennis players aged 12-18. This study employs a three-phase design: first, participants' musical preferences are profiled to create personalized music sequences; second, their mental performance is evaluated through pre- and post-intervention questionnaires measuring perception of success, emotional state, emotion regulation, and flow, with a 45-minute training session followed by a music-accompanied exercise; and third, physical performance is assessed using a battery of tests for muscular strength, endurance, agility, and flexibility, conducted both with and without music to determine its impact.
  Data collection will be done using a questionnaire that has been developed based on the literature.

SUMMARY:
Optimal athletic performance is the result of a synergy between physical abilities and mental skills. Faced with increasing pressure in the world of tennis, athletes are constantly seeking new methods to optimize their performance. Music is a non-pharmacological tool that has demonstrated its effectiveness in reducing anxiety and improving sports performance. This innovative study explores the use of music as a tool to enhance the physical and mental abilities of young Tunisian tennis players. The results of this research could revolutionize training practices and offer new tools to help athletes reach their full potential.

Work objectives: Evaluate the impact of a musical intervention on the physical and mental performance of athletes, particularly young tennis players.

ELIGIBILITY:
Inclusion Criteria:

* Competitive category : Participants must be regular tennis players (number of hours per week) who engage in organized tennis activities (e.g., regular training or participation in competitions).
* Agreement to participate: Participants (players and/or their legal representatives) who agree to participate in the study.

Exclusion Criteria:

* Player's age <10 and > 18 years.
* Non-regular young tennis players (Recreational category): Participants who do not engage in tennis practice regularly.
* Diagnosed psychiatric disorder
* Hearing disorder Severe hearing impairments and certain types of tinnitus. Severe neurological disorders: auditory epilepsy and musicogenic epilepsy (audiogenic seizures are a rare neurological condition characterized by seizures triggered by auditory stimulation).

Amusia and musical deafness (a neurological anomaly where rhythm, melody, and musical chords are not perceived).

Specific psychological issues. Personal sensitivities to certain types of music. History of trauma related to music (intense emotional reactions to certain types of music).

* Refusal to participate: Participants (players and/or their legal epresentatives) who refuse to participate in the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The Perception of Success Questionnaire | before and immediately after intervention
  Perception of Success Questionnaire was designed to measure goal orientation. It is one of the most frequently cited questionnaires on motivation in sport A, B : Strongly agree, C : neutral , D,E : strongly disagree

CONTACTS AND LOCATIONS:
Locations (1):
- TUN, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided